CLINICAL TRIAL: NCT00930787
Title: A Multicenter, Prospective, Randomized, Controlled, Single-Blinded Study of Strattice Reconstructive Tissue Matrix vs Proceed
Brief Title: Hernia Repair in Multiply Morbid Patients
Acronym: RAM2P
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped early
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LFC2007.03.01
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Ventral Hernia
Keywords: hernia repair, surgical mesh, co-morbidities
MeSH Terms: conditions — Hernia, Ventral | interventions — Herniorrhaphy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strattice Reconstructive Tissue Matrix (Experimental): Use of Strattice Reconstructive Tissue Matrix to support hernia repair
  Interventions: Device: Strattice Reconstructive Tissue Matrix (Hernia Repair)
- Proceed Surgical Mesh (Active Comparator): Use of Proceed Surgical Mesh to support hernia repair
  Interventions: Device: Proceed Surgical Mesh (Hernia repair)

INTERVENTIONS:
Device: Strattice Reconstructive Tissue Matrix (Hernia Repair) — Hernia repair will be performed, in an open fashion and defect will be closed or reduced in size using musculofascial centralization procedures to reestablish midline.
  Arms: Strattice Reconstructive Tissue Matrix
Device: Proceed Surgical Mesh (Hernia repair) — Hernia repair will be performed, in an open fashion and defect will be closed or reduced in size using musculofascial centralization procedures to reestablish midline.
  Arms: Proceed Surgical Mesh

SUMMARY:
Support of a ventral hernia repair with a prosthetic mesh has been demonstrated to result in a diminished rate of hernia recurrence. The patient with co-morbidities undergoing hernia repair is at increased risk of wound related complications, which may be exacerbated by the choice of prosthetic mesh, and which are known to influence the ultimate rate of hernia recurrence. It is hypothesized that patients receiving a mesh of biologic origin may experience fewer wound related complications and hence at least an equal rate of hernia recurrence, compared to those receiving a synthetic mesh.

ELIGIBILITY:
Inclusion Criteria:

* Adults of either gender
* must have 2 or more co-morbidities

Exclusion Criteria:

* local or systemic infection
* expected survival of <24 months
* non-ambulatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martindale, MD, Principal Investigator — Oregon Health and Science University
Locations (13):
- United States (13):
  - Louisiana Status University Health Sciences Center, New Orleans, Louisiana
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Boston Veterans Administration Healthcare System, West Roxbury, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Truman Medical Center, Kansas City, Missouri
  - Long Island Jewish - North Shore, Lake Success, New York
  - University Hospital - Case Western, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Scott & White Medical Center, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 subjects recruited from 9 US sites between August 2009 and May 2010.
Period: Overall Study
Arm/Group | Strattice Reconstructive Tissue Matrix | Proceed Surgical Mesh
Started | 14 | 9
Completed | 14 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strattice Reconstructive Tissue Matrix | Proceed Surgical Mesh | Total
Number analyzed (Participants) | 14 | 9 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.47) | 52.7 (13.54) | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Surgical Site Events (SSEs)
Time Frame: Postoperative Day 30
Population: Study was terminated early and no analyses were conducted.
Arm/Group | Strattice Reconstructive Tissue Matrix | Proceed Surgical Mesh
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Strattice Reconstructive Tissue Matrix | Proceed Surgical Mesh
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/9
Other Adverse Events (participants affected / at risk) | 14/14 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strattice Reconstructive Tissue Matrix (N=14) | Proceed Surgical Mesh (N=9)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strattice Reconstructive Tissue Matrix (N=14) | Proceed Surgical Mesh (N=9)
Incisional drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 4 (5) | 1 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localised intraabdominal fluid (Gastrointestinal disorders) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 3 (5) | 2 (5)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 4 (4) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (3)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No